CLINICAL TRIAL: NCT05078242
Title: Virtual Reality - Chronic Pain At-Home Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-13471
Record Dates: First submitted 2021-10-12; First posted 2021-10-14 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: EaseVRx sessions (Experimental): This is a study of patients with chronic pain to assess usability of a VR device at home. The main goals are 1) to collect data on feasibility of recruitment, 2) to collect data on daily adherence to therapy, and 3) to collect preliminary effectiveness data on pain and mood outcomes. There will be 7 sessions over one week, with each session lasting about 2-16 minutes. All patients recruited will be in the active arm; this is not a randomized pilot study.
  Interventions: Device: EaseVRx

INTERVENTIONS:
Device: EaseVRx — Participants will experience 7 sessions of the EaseVRx device for chronic pain.

SUMMARY:
This is a short pilot usability study of a virtual reality device for patients with chronic pain.

DETAILED DESCRIPTION:
The investigators will conduct a study of patients with chronic pain to collect feasibility of recruitment data, adherence to therapy data, and preliminary effectiveness data. All patients will be in the active arm, this is not a randomized study.

The intervention being piloted is the EaseVRx (AppliedVR, Los Angeles, CA) VR hardware and software. EaseVRx incorporates evidence-based principles of cognitive behavioral therapy, mindfulness, and pain neuroscience education into an immersive and enhanced biofeedback experience. EaseVRx includes breathing training and relaxation response exercises that activate the parasympathetic nervous system. EaseVRx was designed for at-home use and comes with a sequence of daily immersive experiences. Each session will include one VR experience, which is 2-16 minutes in length (average of 6 minutes). This study will last one week, or 7 total sessions (out of 56 total sessions).

Participants will complete one survey at 3 days over the telephone assessing pain, mood, adherence to the device, and overall satisfaction. Then participants will complete an additional assessment when the device is returned after day 7, again assessing pain, mood, overall adherence to the device, and overall satisfaction.

The investigators are recruiting participants from the VR Usability Study (IRB # 2021-13108) who expressed interest in participating in further research. As this is a pilot feasibility trial, the plan is to recruit between 5 and 10 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Chronic pain (using self-report) with pain intensity >=4 and confirmed by ICD-10 codes in medical record
3. Fluency in English

Exclusion Criteria:

1. Inability to give informed consent
2. Current or prior diagnosis of epilepsy, seizure disorder, dementia, migraines
3. Medical condition predisposing to nausea or dizziness
4. Hypersensitivity to flashing light or motion
5. No stereoscopic vision or severe hearing impairment
6. Injury to eyes, face, or neck that prevents use of VR headset
7. Currently pregnant, by self-report

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
% of participants contacted that are enrolled | at study 1 day visit
  The investigators will determine feasibility by measuring the % of participants that are contacted who are enrolled.

SECONDARY OUTCOMES:
Satisfaction with VR experience | at study 1 day visit
  The investigators will use the Global Impression of Change Scale, which is a 7 point Likert type scale, at the conclusion of the VR experience to measure patient's perceived impression of change before and after VR.
Change in Mood | at study 1 day visit
  The investigators will use the Brief Mood Introspection Scale, a 16-item scale, to measure change in mood before and after VR
Change in Pain Intensity | at study 1 day visit
  The investigators will use a 1-item pain intensity score (0-10) both before and after VR

CONTACTS AND LOCATIONS:
Overall Officials: Hector Perez, MS, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States